CLINICAL TRIAL: NCT02331264
Title: Cardiac Assessment of Patients With Hip Implants
Status: Completed | Type: Observational
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Professor Alister Hart, Professor Alister Hart, Professor of Orthopaedic Surgery, Director of Research and Development, Royal National Orthopaedic Hospital NHS Trust
Other Study IDs: 157144
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Cardiomyopathy; Cardiac Failure
Keywords: Cardiac Toxicity; Metal on Metal Hip Implants
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MoM >7ppb: Patients with Metal on Metal hip implants and blood metal ions above the Medicines and Healthcare Products Regulatory Agency (MHRA) threshold of 7 parts per billion
  Interventions: Other: Exposure to metal debris
- MoM <7ppb: Patients with Metal on Metal hip implants and blood metal ions below the MHRA threshold of 7 parts per billion
- Non MoM: Patients with non Metal bearing hip implants such as Ceramic on Ceramic or Plastic

INTERVENTIONS:
Other: Exposure to metal debris — The 3 groups are defined by the patients exposure to metal debris from a hip implant. This is either elevated metal ions in those with poorly functioning metal on metal hip implants, or low metal ion levels in those with well functioning metal hip implants, and a second control group of patients with non melt bearing hip implants.
  Groups: MoM >7ppb

SUMMARY:
PRIMARY OBJECTIVE To establish the effect of metal ion release from metal hip implants on cardiac function

STUDY OUTCOME MEASURES

To assess the effect of metal ions from hip implants on cardiac function as measured by Cardiac Magnetic Resonance Imaging (CMR) and Echocardiogram. This involves the surrogate detection of cobalt ion deposition within cardiac tissues and assessment of ejection fraction and tissue characterization (with and without contrast).

STUDY IMPACT

With 60,000 patients having a metal on metal (MOM) hip implant in the United Kingdom (UK), and over a million worldwide, there is need to clarify this important question, which is the source of significant concern amongst patients and surgeons alike. Also, this problem is not unique to MOM hips since all hip implants contain metal and as seen in various case reports high blood cobalt levels have arisen after catastrophic failure (e.g. fracture of a ceramic bearing surface) leading to abnormal wear of the implant and release of metal ions into the body. In the UK, over 80,000 hip implants are inserted annually.

DETAILED DESCRIPTION:
BACKGROUND

Metal-on-metal (MOM) hip implants have a risk of releasing metal ions upon wear of the component material. Some of the metal ions (e.g. cobalt and chromium) from the metal implant or from the metal particles will enter the bloodstream.

The Food and Drug Administration (FDA, USA) recently highlighted systemic toxicity from metal on metal hip implants as a cause for concern and recommended that patients with systemic symptoms are assessed with a particular focus on cardiovascular, neurological, endocrinological (especially thyroid), and renal systems.

A number of cases of suspected toxicity to circulating cobalt and chromium from MOM hip implants, including cardiac toxicity, have been reported recently. The most profound case involves a patient who died from cardiac failure secondary to cardiomyopathy and cobalt deposition within the cardiac tissues. A recent cross sectional health screen and isolated case reports, suggest that raised metal ion levels have the potential to cause cardiomyopathy and cardiac failure. Such cases have raised public anxiety in the process.

Blood metal ions released from metal hip implants are increasingly recognized as a potential cause of local and distant abnormal tissue responses, since cobalt and chromium is released into the peri-prosthetic tissues and transported systemically throughout the body. Component design and positioning are associated with increased wear and as a result raised metal ion levels. However, a definitive causal link to systemic symptoms still remains to be established.

Iron overload disorders affecting the heart or liver is a significant cause of morbidity in primary and secondary haemochromatosis and thalassaemia. Excessive iron deposition within cardiac tissues can lead to premature death secondary to fatal arrhythmias and heart failure. Cardiovascular magnetic resonance (CMR) imaging has revolutionised the management of this particular group of patients by allowing a robust non-invasive method of detecting iron loading.

CMR is the gold-standard method of assessing cardiac volumes, function and mass. It's unique strength over other imaging modalities is tissue characterization with and without the use of contrast agents. Myocardial iron is detected due to the effects on relaxation times through the interaction of iron with hydrogen nuclei in normal cardiac tissue. Cobalt is a ferromagnetic metal containing unpaired electrons allowing it to align in parallel to applied magnetic fields, and therefore should be detected by MRI in a similar way to iron.

RATIONALE

No study has attempted to identify cobalt deposition within cardiac tissue using cardiac MRI. We therefore aim to detect cobalt deposition in the cardiac tissue of patients with metal hip implants and markedly raised cobalt blood ion levels. If detected, we aim to assess whether this had any clinical effect on cardiac function.

Our hypothesis is that there is no discernable effect on cardiac function detectable on Cardiac MRI and Echocardiography in patients with raised blood cobalt ion levels.

Case Controlled Cohort Observation study

Three groups of patients will be identified with Hip implants (matched for age, sex and time since surgery).

1. Patients with MOM hip implant and raised metal ion level (>7ppb) - N=30
2. Patients with MOM hip implant and Normal Metal ion level (<7ppb) - N=30
3. Patients with non-metal bearing hip implant (Ceramic on Ceramic/Polyethylene (COC/COP)) - N=30

Selection into each group will be defined by metal ion blood tests and hip implant type. Patients with two consecutive blood tests at the appropriate level and less than 10% variation (in the last 12 months) will be included, or those with a blood test at the appropriate level taken in the last 3 months will be included.

The cardiologist will be blinded with regards to patient grouping, to ensure there is no bias when reporting the clinical and cardiological investigations results in light of the presence or absence of raised blood metal ions.

All participants enrolled will:

* Be assessed by a cardiologist
* Have a cardiac MRI, an ECHOcardiogram, and an Electrocardiogram (ECG)

These clinical data will be analysed and compared to assess if a significant difference exists between the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years of age
2. Either male or female
3. Metal on Metal hip implant (ceramic on ceramic hip implant for patients within control group)
4. Implanted greater than 12 months (i.e. beyond the bedding in period of the implant)
5. Suitable for MRI scanning (no contraindications for Magnetic scanning - for instance metal implants in eyes/brain/heart, and claustrophobia)
6. Consenting to the proposed research activity

Exclusion Criteria:

1. Age below 18 years
2. Metal hip implant not considered as MOM or Ceramic on Ceramic (COC) if part of the control group
3. Not suitable to undergo MRI scanning (contra-indications or claustrophobia)
4. Revised hip implant
5. Atrial Fibrillation
6. Poor renal function (eGFR<30)
7. Consent not given
8. Vulnerable adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hip replacements. Groups 1 and 2 include patients with Metal on Metal hip replacements. Group 3 includes patients with non Metal bearing hip replacements including Ceramic on Ceramic Hip replacements.
  All three groups will be matched for Age, Sex, Time since hip Implantation, and diabetes status.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Cardiac Ejection Fraction | 1 hour
  Use of Echocardiogram and Cardiac MRI (Gold Standard) for assessment of ejection fraction of the heart

SECONDARY OUTCOMES:
Detection of Cobalt Metal Ion deposition within cardiac tissues | 30 mins
  Use of Cardiac MRI series T1 and T2* relaxation times, which correlate with metal debris within cardiac tissues

CONTACTS AND LOCATIONS:
Overall Officials: Alister Hart, MD,FRCSG, Principal Investigator — Professor of Orthopaedic Surgery at UCL and Consultant Orthopaedic Surgeon at the RNOH. Director of research and development at the RNOH.
Locations (2):
- United Kingdom (2):
  - The Heart Hospital, London, London
  - Royal National Orthopaedic Hospital, Stanmore, London

IPD SHARING:
Plan to Share IPD: Yes
publication submitted

REFERENCES:
- [Result] Steens W, von Foerster G, Katzer A. Severe cobalt poisoning with loss of sight after ceramic-metal pairing in a hip--a case report. Acta Orthop. 2006 Oct;77(5):830-2. doi: 10.1080/17453670610013079. No abstract available. PMID 17068719
- [Result] Rizzetti MC, Liberini P, Zarattini G, Catalani S, Pazzaglia U, Apostoli P, Padovani A. Loss of sight and sound. Could it be the hip? Lancet. 2009 Mar 21;373(9668):1052. doi: 10.1016/S0140-6736(09)60490-6. No abstract available. PMID 19304018
- [Result] Ikeda T, Takahashi K, Kabata T, Sakagoshi D, Tomita K, Yamada M. Polyneuropathy caused by cobalt-chromium metallosis after total hip replacement. Muscle Nerve. 2010 Jul;42(1):140-3. doi: 10.1002/mus.21638. PMID 20544916
- [Result] Oldenburg M, Wegner R, Baur X. Severe cobalt intoxication due to prosthesis wear in repeated total hip arthroplasty. J Arthroplasty. 2009 Aug;24(5):825.e15-20. doi: 10.1016/j.arth.2008.07.017. Epub 2008 Oct 2. PMID 18835128
- [Result] Tower SS. Arthroprosthetic cobaltism: neurological and cardiac manifestations in two patients with metal-on-metal arthroplasty: a case report. J Bone Joint Surg Am. 2010 Dec 1;92(17):2847-51. doi: 10.2106/JBJS.J.00125. Epub 2010 Oct 29. No abstract available. PMID 21037026
- [Result] Tower SS. Arthroprosthetic cobaltism associated with metal on metal hip implants. BMJ. 2012 Jan 17;344:e430. doi: 10.1136/bmj.e430. No abstract available. PMID 22252702
- [Result] Mao X, Wong AA, Crawford RW. Cobalt toxicity--an emerging clinical problem in patients with metal-on-metal hip prostheses? Med J Aust. 2011 Jun 20;194(12):649-51. doi: 10.5694/j.1326-5377.2011.tb03151.x. PMID 21692725
- [Result] Gilbert CJ, Cheung A, Butany J, Zywiel MG, Syed K, McDonald M, Wong F, Overgaard C. Hip pain and heart failure: the missing link. Can J Cardiol. 2013 May;29(5):639.e1-2. doi: 10.1016/j.cjca.2012.10.015. Epub 2013 Jan 9. PMID 23313008
- [Result] Prentice JR, Clark MJ, Hoggard N, Morton AC, Tooth C, Paley MN, Stockley I, Hadjivassiliou M, Wilkinson JM. Metal-on-metal hip prostheses and systemic health: a cross-sectional association study 8 years after implantation. PLoS One. 2013 Jun 10;8(6):e66186. doi: 10.1371/journal.pone.0066186. Print 2013. PMID 23762480
- [Result] Machado C, Appelbe A, Wood R. Arthroprosthetic cobaltism and cardiomyopathy. Heart Lung Circ. 2012 Nov;21(11):759-60. doi: 10.1016/j.hlc.2012.03.013. Epub 2012 Apr 18. PMID 22520206
- [Result] Cohen D. How safe are metal-on-metal hip implants? BMJ. 2012 Feb 28;344:e1410. doi: 10.1136/bmj.e1410. No abstract available. PMID 22374741
- [Result] Jacobs JJ, Skipor AK, Patterson LM, Hallab NJ, Paprosky WG, Black J, Galante JO. Metal release in patients who have had a primary total hip arthroplasty. A prospective, controlled, longitudinal study. J Bone Joint Surg Am. 1998 Oct;80(10):1447-58. doi: 10.2106/00004623-199810000-00006. PMID 9801213
- [Result] Case CP, Langkamer VG, James C, Palmer MR, Kemp AJ, Heap PF, Solomon L. Widespread dissemination of metal debris from implants. J Bone Joint Surg Br. 1994 Sep;76(5):701-12. PMID 8083255
- [Result] Merritt K, Brown SA. Release of hexavalent chromium from corrosion of stainless steel and cobalt-chromium alloys. J Biomed Mater Res. 1995 May;29(5):627-33. doi: 10.1002/jbm.820290510. PMID 7622548
- [Result] De Haan R, Pattyn C, Gill HS, Murray DW, Campbell PA, De Smet K. Correlation between inclination of the acetabular component and metal ion levels in metal-on-metal hip resurfacing replacement. J Bone Joint Surg Br. 2008 Oct;90(10):1291-7. doi: 10.1302/0301-620X.90B10.20533. PMID 18827237
- [Result] Langton DJ, Sprowson AP, Joyce TJ, Reed M, Carluke I, Partington P, Nargol AV. Blood metal ion concentrations after hip resurfacing arthroplasty: a comparative study of articular surface replacement and Birmingham Hip Resurfacing arthroplasties. J Bone Joint Surg Br. 2009 Oct;91(10):1287-95. doi: 10.1302/0301-620X.91B10.22308. PMID 19794161
- [Result] Langton DJ, Jameson SS, Joyce TJ, Webb J, Nargol AV. The effect of component size and orientation on the concentrations of metal ions after resurfacing arthroplasty of the hip. J Bone Joint Surg Br. 2008 Sep;90(9):1143-51. doi: 10.1302/0301-620X.90B9.20785. PMID 18757952
- [Result] Hart AJ, Skinner JA, Henckel J, Sampson B, Gordon F. Insufficient acetabular version increases blood metal ion levels after metal-on-metal hip resurfacing. Clin Orthop Relat Res. 2011 Sep;469(9):2590-7. doi: 10.1007/s11999-011-1930-y. Epub 2011 Jun 9. PMID 21656317
- [Result] Matthies AK, Henckel J, Cro S, Suarez A, Noble PC, Skinner J, Hart AJ. Predicting wear and blood metal ion levels in metal-on-metal hip resurfacing. J Orthop Res. 2014 Jan;32(1):167-74. doi: 10.1002/jor.22459. Epub 2013 Sep 21. PMID 24115200
- [Result] Devlin JJ, Pomerleau AC, Brent J, Morgan BW, Deitchman S, Schwartz M. Clinical features, testing, and management of patients with suspected prosthetic hip-associated cobalt toxicity: a systematic review of cases. J Med Toxicol. 2013 Dec;9(4):405-15. doi: 10.1007/s13181-013-0320-0. PMID 24222555
- [Result] Baur LH. Early detection of iron overload in the heart: a key role for MRI! Int J Cardiovasc Imaging. 2009 Dec;25(8):789-90. doi: 10.1007/s10554-009-9538-y. Epub 2009 Nov 24. No abstract available. PMID 19937124
- [Result] Chu WC, Au WY, Lam WW. MRI of cardiac iron overload. J Magn Reson Imaging. 2012 Nov;36(5):1052-9. doi: 10.1002/jmri.23628. PMID 23090916
- [Result] Gulati V, Harikrishnan P, Palaniswamy C, Aronow WS, Jain D, Frishman WH. Cardiac involvement in hemochromatosis. Cardiol Rev. 2014 Mar-Apr;22(2):56-68. doi: 10.1097/CRD.0b013e3182a67805. PMID 24503941
- [Result] Pepe A, Positano V, Santarelli MF, Sorrentino F, Cracolici E, De Marchi D, Maggio A, Midiri M, Landini L, Lombardi M. Multislice multiecho T2* cardiovascular magnetic resonance for detection of the heterogeneous distribution of myocardial iron overload. J Magn Reson Imaging. 2006 May;23(5):662-8. doi: 10.1002/jmri.20566. PMID 16568436
- [Result] Anderson LJ, Holden S, Davis B, Prescott E, Charrier CC, Bunce NH, Firmin DN, Wonke B, Porter J, Walker JM, Pennell DJ. Cardiovascular T2-star (T2*) magnetic resonance for the early diagnosis of myocardial iron overload. Eur Heart J. 2001 Dec;22(23):2171-9. doi: 10.1053/euhj.2001.2822. PMID 11913479
- [Result] Hundley WG, Bluemke D, Bogaert JG, Friedrich MG, Higgins CB, Lawson MA, McConnell MV, Raman SV, van Rossum AC, Flamm S, Kramer CM, Nagel E, Neubauer S. Society for Cardiovascular Magnetic Resonance guidelines for reporting cardiovascular magnetic resonance examinations. J Cardiovasc Magn Reson. 2009 Mar 3;11(1):5. doi: 10.1186/1532-429X-11-5. PMID 19257889
- [Result] Kramer CM, Barkhausen J, Flamm SD, Kim RJ, Nagel E; Society for Cardiovascular Magnetic Resonance Board of Trustees Task Force on Standardized Protocols. Standardized cardiovascular magnetic resonance (CMR) protocols 2013 update. J Cardiovasc Magn Reson. 2013 Oct 8;15(1):91. doi: 10.1186/1532-429X-15-91. PMID 24103764
- [Result] Quarta G, Sado DM, Moon JC. Cardiomyopathies: focus on cardiovascular magnetic resonance. Br J Radiol. 2011 Dec;84 Spec No 3(Spec Iss 3):S296-305. doi: 10.1259/bjr/67212179. PMID 22723536
- [Result] Hart AJ, Satchithananda K, Liddle AD, Sabah SA, McRobbie D, Henckel J, Cobb JP, Skinner JA, Mitchell AW. Pseudotumors in association with well-functioning metal-on-metal hip prostheses: a case-control study using three-dimensional computed tomography and magnetic resonance imaging. J Bone Joint Surg Am. 2012 Feb 15;94(4):317-25. doi: 10.2106/JBJS.J.01508. PMID 22336970
- [Result] Hart AJ, Sabah S, Henckel J, Lewis A, Cobb J, Sampson B, Mitchell A, Skinner JA. The painful metal-on-metal hip resurfacing. J Bone Joint Surg Br. 2009 Jun;91(6):738-44. doi: 10.1302/0301-620X.91B6.21682. PMID 19483225
- [Result] Hart AJ, Sabah SA, Bandi AS, Maggiore P, Tarassoli P, Sampson B, A Skinner J. Sensitivity and specificity of blood cobalt and chromium metal ions for predicting failure of metal-on-metal hip replacement. J Bone Joint Surg Br. 2011 Oct;93(10):1308-13. doi: 10.1302/0301-620X.93B10.26249. PMID 21969427
- [Result] Back DL, Young DA, Shimmin AJ. How do serum cobalt and chromium levels change after metal-on-metal hip resurfacing? Clin Orthop Relat Res. 2005 Sep;438:177-81. doi: 10.1097/01.blo.0000166901.84323.5d. PMID 16131888
- [Result] Ball ST, Severns D, Linn M, Meyer RS, Swenson FC. What happens to serum metal ion levels after a metal-on-metal bearing is removed? J Arthroplasty. 2013 Sep;28(8 Suppl):53-5. doi: 10.1016/j.arth.2013.06.040. Epub 2013 Aug 12. PMID 23948123
- [Result] Ebreo D, Khan A, El-Meligy M, Armstrong C, Peter V. Metal ion levels decrease after revision for metallosis arising from large-diameter metal-on-metal hip arthroplasty. Acta Orthop Belg. 2011 Dec;77(6):777-81. PMID 22308623
- [Result] Newton AW, Ranganath L, Armstrong C, Peter V, Roberts NB. Differential distribution of cobalt, chromium, and nickel between whole blood, plasma and urine in patients after metal-on-metal (MoM) hip arthroplasty. J Orthop Res. 2012 Oct;30(10):1640-6. doi: 10.1002/jor.22107. Epub 2012 Mar 23. PMID 22447496
- [Result] Urban RM, Jacobs JJ, Tomlinson MJ, Gavrilovic J, Black J, Peoc'h M. Dissemination of wear particles to the liver, spleen, and abdominal lymph nodes of patients with hip or knee replacement. J Bone Joint Surg Am. 2000 Apr;82(4):457-76. doi: 10.2106/00004623-200004000-00002. PMID 10761937
- [Result] Afolaranmi GA, Akbar M, Brewer J, Grant MH. Distribution of metal released from cobalt-chromium alloy orthopaedic wear particles implanted into air pouches in mice. J Biomed Mater Res A. 2012 Jun;100(6):1529-38. doi: 10.1002/jbm.a.34091. Epub 2012 Mar 15. PMID 22419548
- [Result] Pelclova D, Sklensky M, Janicek P, Lach K. Severe cobalt intoxication following hip replacement revision: clinical features and outcome. Clin Toxicol (Phila). 2012 Apr;50(4):262-5. doi: 10.3109/15563650.2012.670244. PMID 22455358
- [Result] Zywiel MG, Brandt JM, Overgaard CB, Cheung AC, Turgeon TR, Syed KA. Fatal cardiomyopathy after revision total hip replacement for fracture of a ceramic liner. Bone Joint J. 2013 Jan;95-B(1):31-7. doi: 10.1302/0301-620X.95B1.30060. PMID 23307670
- [Result] van Lingen CP, Ettema HB, Timmer JR, de Jong G, Verheyen CC. Clinical manifestations in ten patients with asymptomatic metal-on-metal hip arthroplasty with very high cobalt levels. Hip Int. 2013 Sep-Oct;23(5):441-4. doi: 10.5301/hipint.5000054. Epub 2013 Jun 28. PMID 23813157
- [Result] Alexander CS. Cobalt-beer cardiomyopathy. A clinical and pathologic study of twenty-eight cases. Am J Med. 1972 Oct;53(4):395-417. doi: 10.1016/0002-9343(72)90136-2. No abstract available. PMID 4263183
- [Result] Linna A, Oksa P, Groundstroem K, Halkosaari M, Palmroos P, Huikko S, Uitti J. Exposure to cobalt in the production of cobalt and cobalt compounds and its effect on the heart. Occup Environ Med. 2004 Nov;61(11):877-85. doi: 10.1136/oem.2003.009605. PMID 15477280
- [Result] CARTWRIGHT GE. The relationship of copper, cobalt, and other trace elements to hemopoiesis. Am J Clin Nutr. 1955 Jan-Feb;3(1):11-9. doi: 10.1093/ajcn/3.1.11. No abstract available. PMID 14349898
- [Result] Brock T, Stopford W. Bioaccessibility of metals in human health risk assessment: evaluating risk from exposure to cobalt compounds. J Environ Monit. 2003 Aug;5(4):71N-76N. doi: 10.1039/b307520f. No abstract available. PMID 12948221
- [Result] KRISS JP, CARNES WH, GROSS RT. Hypothyroidism and thyroid hyperplasia in patients treated with cobalt. J Am Med Assoc. 1955 Jan 8;157(2):117-21. doi: 10.1001/jama.1955.02950190017004. No abstract available. PMID 13211322
- [Result] Hallab N, Merritt K, Jacobs JJ. Metal sensitivity in patients with orthopaedic implants. J Bone Joint Surg Am. 2001 Mar;83(3):428-36. doi: 10.2106/00004623-200103000-00017. PMID 11263649
- [Result] Hallab NJ. Lymphocyte transformation testing for quantifying metal-implant-related hypersensitivity responses. Dermatitis. 2004 Jun;15(2):82-90. doi: 10.2310/6620.2004.03054. PMID 15473335
- [Result] Atanaskova Mesinkovska N, Tellez A, Molina L, Honari G, Sood A, Barsoum W, Taylor JS. The effect of patch testing on surgical practices and outcomes in orthopedic patients with metal implants. Arch Dermatol. 2012 Jun;148(6):687-93. doi: 10.1001/archdermatol.2011.2561. PMID 22351785
- [Result] Leikin JB, Karydes HC, Whiteley PM, Wills BK, Cumpston KL, Jacobs JJ. Outpatient toxicology clinic experience of patients with hip implants. Clin Toxicol (Phila). 2013 May;51(4):230-6. doi: 10.3109/15563650.2013.768343. Epub 2013 Feb 20. PMID 23421810